CLINICAL TRIAL: NCT01455272
Title: Clinical Study of Granulocyte Colony-stimulating Factor (G-CSF)-Primed, Peripheral-blood Progenitor Cells for the Prevention of Relapse Advanced Stage Leukemia
Brief Title: New Therapy for Advanced Stage Leukemia After Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, director of Peking University People's Hospital，Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PUPH IRB [2010] (78)
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high-risk leukemia (Experimental)
  Interventions: Procedure: prophylactic GPBPCI

INTERVENTIONS:
Procedure: prophylactic GPBPCI — A G-CSF-primed PBPCI was planned within day 60 post-transplantation before hematologic relapse was diagnosed
  Other Names: modified DLI

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is one of the best, and sometimes the only, option for the treatment of leukemia, particularly for patients with advanced-stage leukemia. However, relapse rate was still very high for advanced-stage leukemia.

It was found in our previous study that infusion of granulocyte colony-stimulating factor (G-CSF)-primed peripheral blood progenitor cells (GPBPC) instead of non-primed lymphocytes exhibited a comparative or stronger graft-versus-leukemia (GVL) effect and comparative or less incidence of GVHD, rarely being complicated with pancytopenia. When GPBPC infusion was combined with the use of short-term immunosuppressant for GVHD prophylaxis, the incidence of fatal GVHD complicated with GPBPCI was further reduced. Our primary data showed the GPBPCI combined with the use of short-term immunosuppressant was feasible in patients with advanced leukemia to prevent relapse after HLA-mismatched HSCT.

The study hypothesis:

Prevention of relapse using granulocyte colony-stimulating factor-primed peripheral blood progenitor cells following hematopoietic stem cell transplantation in patients with advanced-stage acute leukemia can

* reduce relapse rate
* improve survival

DETAILED DESCRIPTION:
A G-CSF-primed PBPCI was planned within day 60 post-transplantation before hematologic relapse was diagnosed in patients for which no GVHD occurred or free of GVHD after 2 weeks off immunosuppression for patients receiving GPBPCI after day 90 post HSCT. Before administration of GPBPCI, serious infection had to be cleared and no serious organ failure could be present. The GPBPCI regimen was comprised of G-CSF-primed PBSCs instead of harvested non-primed donor lymphocytes and short-term immunosuppressive agents for prevention of GVHD after GPBPCI. Chimerism status was examined before and after prophylactic treatment with GPBPCI.

ELIGIBILITY:
Inclusion Criteria:

* high-risk leukemia after HSCT

Exclusion Criteria:

* active GVHD
* early relapse

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
relapse rate | one year after HSCT

SECONDARY OUTCOMES:
survival probability | one year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: XiaoJun Huang, M.D., Principal Investigator — Peking University People's Hospital，Institute of Hematology
Locations (6):
- China (6):
  - Lanzhou General Hospital of Lanzhou Command, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Peking University People's Hospital，Institute of Hematology, Beijing
  - Xinqiao Hospital,Third Military Medical University, Chongqing

REFERENCES:
- [Derived] Yan CH, Wang Y, Sun YQ, Cheng YF, Mo XD, Wang FR, Chen YH, Zhang YY, Han TT, Chen H, Xu LP, Zhang XH, Liu KY, Huang XJ. Optimized therapeutic strategy for patients with refractory or relapsed acute myeloid leukemia: long-term clinical outcomes and health-related quality of life assessment. Cancer Commun (Lond). 2022 Dec;42(12):1387-1402. doi: 10.1002/cac2.12376. Epub 2022 Oct 23. PMID 36274263
- [Derived] Zhou YL, Wu LX, Peter Gale R, Wang ZL, Li JL, Jiang H, Jiang Q, Jiang B, Cao SB, Lou F, Sun Y, Wang CC, Liu YR, Wang Y, Chang YJ, Xu LP, Zhang XH, Liu KY, Ruan GR, Huang XJ. Mutation topography and risk stratification for de novo acute myeloid leukaemia with normal cytogenetics and no nucleophosmin 1 (NPM1) mutation or Fms-like tyrosine kinase 3 internal tandem duplication (FLT3-ITD). Br J Haematol. 2020 Jul;190(2):274-283. doi: 10.1111/bjh.16526. Epub 2020 Feb 26. PMID 32103499
- [Derived] Yan CH, Liu QF, Wu DP, Zhang X, Xu LP, Zhang XH, Wang Y, Huang H, Bai H, Huang F, Ma X, Huang XJ. Prophylactic Donor Lymphocyte Infusion (DLI) Followed by Minimal Residual Disease and Graft-versus-Host Disease-Guided Multiple DLIs Could Improve Outcomes after Allogeneic Hematopoietic Stem Cell Transplantation in Patients with Refractory/Relapsed Acute Leukemia. Biol Blood Marrow Transplant. 2017 Aug;23(8):1311-1319. doi: 10.1016/j.bbmt.2017.04.028. Epub 2017 May 5. PMID 28483716